CLINICAL TRIAL: NCT06781151
Title: A Real-world Study to Explore Personalized Treatment for Patients With Recurrent Gynecological Malignancies Based on Molecular Profiling and Multidisciplinary Team Consultation
Brief Title: A Study to Explore Personalized Treatment for Patients With Recurrent Gynecological Malignancies Based on MTB
Acronym: RWS-MTB
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jihong Liu, professor, Sun Yat-sen University
Other Study IDs: 2023-FXY-274
Record Dates: First submitted 2025-01-05; First posted 2025-01-17 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer Recurrent; Endometrial Cancer Recurrent; Cervical Cancer Recurrent
Keywords: genomic sequencing; molecular tumor boards; recurrent ovarian cancer; recurrent endometrial cancer; recurrent cervical cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional, real-world study divided into two parts: a retrospective study and a prospective study.

The main question it aims to answer is:

Will genomic sequencing and molecular tumor boards lead to clinical responses in patients with recurrent ovarian, cervical, or endometrial cancer? The retrospective arm will analyze data from patients with recurrent gynecological malignancies (ovarian, cervical, or endometrial) who underwent multidisciplinary consultations at our institution from January 2022 onward. Data collected will include tumor tissue genomic sequencing results, medical histories, multidisciplinary consultation recommendations, and subsequent treatment courses. This analysis will examine the implementation and clinical efficacy of personalized targeted therapies guided by molecular tumor profiling and multidisciplinary consultation.

The prospective arm will enroll 200 patients with recurrent gynecological malignancies (ovarian, cervical, or endometrial) referred for multidisciplinary consultation. Tumor tissue and blood samples will undergo next-generation sequencing (NGS) to determine molecular tumor profiles. A multidisciplinary expert panel will formulate individualized treatment strategies based on these profiles, patient clinical data, and treatment history. Attending physicians will determine the final treatment plan, integrating multidisciplinary recommendations with patient preferences, comorbidity considerations, drug toxicity assessments, insurance coverage for off-label medications, and the availability of investigational drug trials. This arm aims to observe and evaluate the clinical efficacy of personalized treatment plans developed through molecular tumor profiling and multidisciplinary consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent ovarian, cervical, or endometrial cancer referred for multidisciplinary consultation by a gynecological oncologist;
* Presence of at least one evaluable lesion;
* Willingness to participate in multidisciplinary consultation;
* Age 18 years or older;
* Sufficient tumor tissue for next-generation sequencing (NGS) with a tumor content greater than 32%;
* Informed consent provided by the participant, indicating understanding of the study procedures and willingness to participate.

Exclusion Criteria:

* Patients with concurrent malignancies;
* Pregnant patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent ovarian, cervical, or endometrial cancer referred for multidisciplinary consultation by a gynecological oncologist
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2027-06-18 (Estimated)

PRIMARY OUTCOMES:
the overall response rate | an assessment was performed at the end of Cycle 2 or Cycle 3 or Cycle 4 (each cycle is 21-28 days) according to the actual situation
  the overall response rate (ORR) by the presence of radiologically assessable disease by cross-sectional CT or MRI imaging and/or by MIBG or PET scans

SECONDARY OUTCOMES:
the progression free survival (PFS) | 2 years
  the time from the start of treatment until the disease progresses or the patient dies from any cause, whichever comes first.
the overall survival (OS) | 2 years
  a measure of the length of time from the start of treatment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, PhD, Principal Investigator — Sun Yat'sen University Cancer Center
Locations (2):
- China (2):
  - Sun Yat'sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences,Shenzhen Center, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No